CLINICAL TRIAL: NCT07364578
Title: Evaluating the Efficacy of Probiotic Supplements on Osteoarthritis Patients
Brief Title: Probiotic Supplements in Osteoarthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, Lecturer of clinical pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Probiotic1
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome assessors were blinded to participant data. the researcher coded patient data before analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): OA patients will receive only standard of care
  Interventions: Drug: Control
- probiotic group (Experimental): OA patients will receive probiotic supplements (2 times daily) added to the standard of care.
  Interventions: Drug: Probiotic Formula

INTERVENTIONS:
Drug: Probiotic Formula — probiotic supplements (lactobacillus, 2 times daily) added to standard of care
  Arms: probiotic group
Drug: Control — standard of care
  Arms: Control group

SUMMARY:
The current study aims to evaluate the effectiveness of adding probiotics to the standard of care in improving OA patient-related outcomes such as pain, stiffness, and physical activity.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a severe progressive chronic arthropathy causing articular remodeling and inflammation of synovial tissue. The disease involves the entire synovial joint, including the cartilage, joint lining, and subchondral bone. OA causes pain, swelling, and stiffness, consequently hindering the patient's ability to perform their main daily activities, which often leads to social isolation and depression. Up till now, there is no cure for OA treatment options target either symptomatic relief (mainly pain) such as acetaminophen, glucosamine, chondroitin sulfate, and non-steroidal anti-inflammatory drugs (NSAIDs) or structure repair.

Probiotics are live and active microorganisms widely known as the gut's beneficial bacteria. They are taken to alter the GI flora and provide health benefits such as achieving optimal digestion and immunological function.

ELIGIBILITY:
Inclusion Criteria:

Patients (both sexes) aged above 18 years who met the American College of Rheumatology (ACR) clinical criteria for KOA [7] and had symptomatic OA of at least one knee (index knee).

Exclusion Criteria:

1. Rheumatoid arthritis or other active generalized inflammatory comorbidities affecting the gastrointestinal tract (IBD, celiac disease)
2. Performed a total knee replacement on the affected knee or the waiting list for joint replacement
3. surgeries (such as gastric bypass) or Other concomitant injuries can override OA symptoms or interfere with physical activity.
4. Malabsorption disorders, systemic organ failure (liver, renal, cardiac)
5. Use corticosteroids with doses above 10 mg/day or Intra-articular injections during the previous 6 months.
6. Recent antibiotic treatment (i.e., <2 months before the beginning of the study).
7. Pregnancy/breastfeeding
8. Participants who smoked more than 10 cigarettes per day were excluded.
9. Immunosuppressive treatment or impaired immune system
10. Chronic or acute diarrhea
11. Blood/plasma donation/transfusion during the 3 months of the study
12. Non-controlled diabetes
13. Allergy with regards to any of the study product ingredients.
14. Post-traumatic OA (e.g., fractures), congenital hip deformities, or degenerative or non-degenerative neurological conditions can alter pain perception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 3 months
  A self-administered measure used in assessing pain, stiffness, and function in OA patients
Visual Analogue Scale (VAS) | 3 months
  A pain rating scale that represents the severity of symptoms from 0 "no symptoms" to 10 "very severe symptoms." The patient marks the line according to his/her perception of their current state.

SECONDARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | 3 months
  a questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Elsayed, Principal Investigator — Beni-Suef University
Locations (1):
- Asmaa Abdelfattah Elsayed, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No